CLINICAL TRIAL: NCT01355120
Title: THE IPI - Multibasket Trial in Advanced Melanoma: Prospective Clinical Phase II Multibasket Study in Melanoma Patients With Advanced Disease (DeCOG MM-PAL11)
Brief Title: THE IPI - Trial in Advanced Melanoma: Melanoma Patients With Advanced Disease
Acronym: DeCOG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. med. Dirk Schadendorf (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Dirk Schadendorf, Professor, University Hospital, Essen
Organization: University Hospital, Essen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DeCOG -MM-PAL11
Record Dates: First submitted 2010-12-29; First posted 2011-05-17 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2014-06

CONDITIONS: Ocular Melanoma
Keywords: advanced ocular melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- a human immunoglobulin (Experimental): Four infusions (i.v.) of 3mg/kg Ipilimumab in week 1, week 4, week 7 and week 10
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab monotherapy 3mg/kg by four infusion every 3 weeks
  Other Names: Yervoy

SUMMARY:
This is an open-label, multi-center, single-arm clinical phase II study to further characterize the efficacy and safety of ipilimumab in patients with or without systemic pretreatment metastatic ocular melanoma.

The DeCOG-MM-PAL11-Trial will be continued only for patients with ocular melanoma because sufficient numbers of cutaneous and mucosal melanoma patients have already been recruited. In order to allow the separate subgroup analysis as planned in the protocol for ocular melanoma it is mandatory to focus the recruitment to this patient population. Only this will guarantee a valid evaluation of all cohorts. Ocular melanoma is defined as melanomas originated from uvea, the choroid, the ciliary body and conjunctiva. (see McCartney ACE "Pathology of ocular melanomas" British Medical Bulltta, 1995, Vol 51, No 3 pp 678-693) The same criteria and treatment procedure as those used before will be applied for the patients with advanced ocular melanoma. Since no treatment standard in those patients does exist, also patients without prior systemic treatment can be included in this study. Therefore, the 5th inclusion criterion has been adapted in order to enrol the eligible patients.

DETAILED DESCRIPTION:
Treatment:

Treatment with the anti-CTLA-4 mAb Ipilimumab monotherapy of each patient in the scope of this trial is defined as induction plus re-induction of eligible patients until 12 months after first receipt of study medication

Induction phase:

Ipilimumab will be applied to melanoma patients according to the protocol of the completed Medarex study MDX-010-20: Ipilimumab by IV infusion, 3 mg/kg, day 1 (Week 1), 22 (Week 4), 43 (Week 7), 64 (Week 10)

Re-induction:

Patients who progress following stable disease of ≥ 3 months duration starting from diagnosis at week 12 tumor assessment or patients who have progressed following an initial response (partial or complete) assessed at week 12 may be offered additional cycles of therapy with the originally assigned treatment regimen until off-treatment criteria are met, provided they meet re-treatment eligibility requirements. No patient will be re-treated if they experience a Grade 3 or higher gastrointestinal or certain other immune-related adverse events (irAE) (refer to section 5.2 and 5.3). No patient with disease progression following the first cycle of study medication will be permitted to be re-treated with study medication.

Examinations:

The disease will be assessed at baseline, after 12 weeks and for patients with stable disease or better responses, thereafter every 12 weeks in the absence of PD with a maximum of one year. Response evaluation will be done according to immune-related response criteria (Wolchok et al., CCR 2009).

All patients who prematurely discontinued treatment due to a drug-related adverse event prior to Week 12 (in the absence of disease progression) will return for all study visits and procedures including Week 12 and, if appropriate, further re-staging assessments. Any patient with documented progression at any scheduled re-staging visit and who will not receive any re-induction will undergo no further re-staging visits.

Follow-up phase:

Survival will be assessed every 3 months after the final dose of Ipilimumab until the end of the follow-up phase for the individual patient. FU phase for each subject is 1 year following first treatment dose. End of study will be at recruitment finished plus 1 year post start of treatment of last patient thus ensuring that 1 year survival rate can be estimated.

Study duration:

End of study is 1 year post LPFV. Recruiting period for the ocular melanoma:

Period of recruiting 12-18 months Enrolment start date (FPI): QIII 2011 Enrolment finish date (LPI): QI 2013 End of study: QI 2014

ELIGIBILITY:
Inclusion Criteria

Patients meeting all of the following criteria will be considered for admission to the trial:

1. Histologically proven ocular melanoma
2. Measurable disease according to RECIST in unresectable stage III-IV
3. Minimum age of 18 years,
4. Able and willing to give valid written inform consent
5. Patients with or without prior systemic treatment for advanced malignant melanoma are eligible .
6. In case of systemic pre-treatment, an interval of at least 28 days since treatment with chemotherapy, biochemotherapy, surgery, radiation, or immunotherapy is mandatory as well as recovery from any clinically significant toxicity experienced during treatment is recommended. Prior treatment must be completed by the time of ipilimumab administration. Palliative radiation therapy outside of the brain or therapeutic radiation to the brain after the patient's condition is stabilized and systemic steroids required for the management of symptoms due to brain metastases is decreased to the lowest fixed dose possible and does not require the 28-day waiting period. Patient must have recovered from any acute toxicity associated with prior therapy.
7. Expected survival of at least six months
8. ECOG Performance Status 0, 1 or 2.
9. Within the last 2 weeks prior to study day 1 the following laboratory parameters, which should be within the ranges specified:

   Lab Parameter Range White blood cells (WBC) >= 2500/mm3 (≥ 1 2.5 x 109/L) Absolute neutrophil count (ANC) >= 1000/mm3 (≥ 1.0 x 109/L) Platelets ≥75.000/mm3 (≥ 75 x 109/L) Hemoglobin ≥ 9 g/dL (≥ 90 g/L; may be transfused) Creatinine <= 2.0 x ULN Bilirubin total <= 2.0 x ULN (excepted patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL) <= 5 x ULN for patients with liver metastases
10. No childbearing potential or negative pregnancy test of women of childbearing potential performed within 7 days prior to the start of treatment.

Women of childbearing potential (WOCP) must be using an effective method of contraception (Pearl-Index < 1, e.g. oral contraceptives, other hormonal contraceptives [vaginal products, skin patches, or implanted or injectable products], or mechanical products such as an intrauterine device or barrier methods [diaphragm, spermicides]) throughout the study and for up to 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized.

No men of fathering potential or men of fathering potential must be using an effective method of contraception to avoid conception throughout the study and for up to 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized.

WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal.

Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential.

WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) at Baseline within 7 days before the start of ipilimumab and at week 12.

Exclusion Criteria

Patients will be excluded from the study for any of the following reasons:

1. The patient requires concomitant therapy with any of the following: IL 2, interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; any other systemic therapy for cancer including any other experimental treatment.
2. The patient requires chronic use of systemic corticosteroids. Systemic steroids for management of symptoms due to brain mets should be avoided if possible or subject should be stable on the lowest clinically effective dose. Topical or inhalational steroids are permitted.
3. Use of any investigational or non-registered product (drug or vaccine) other than the study treatment.
4. Active autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis).
5. Symptomatic CNS metastases (Remark: Asymptomatic stable, untreated or pretreated central nervous system (CNS) metastasis are allowed)
6. Family history of congenital or hereditary immunodeficiency.
7. The patient is known to be positive for Human Immunodeficiency Virus (HIV) or other chronic infections (HBV, HCV) or has another confirmed or suspected immunosuppressive or immunodeficient condition.
8. The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent or to comply with the trial procedures.
9. Lack of availability for clinical follow-up assessments.
10. The patient has concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
11. Other serious illnesses, e.g., serious infections requiring antibiotics or bleeding disorders.
12. Patients with serious intercurrent illness, requiring hospitalization.
13. For female patients: the patient is pregnant or lactating. Women of childbearing potential: Refusal or inability to use effective means of contraception
14. Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
15. Subjects with melanoma who have another active, concurrent, malignant disease are not eligible for this trial, with the exception of adequately treated basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix.
16. Previous treatment with ipilimumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | alive 12 months after date from the first study drug adminstration
  Overall survival rate at 12 months defined as the rate of patients alive 12 months after the date from the first study treatment for complete study

SECONDARY OUTCOMES:
safety and efficacy parameters | 12 months after date from the first study drug adminstration
  The primary endpoint is the one-year survival rate. It is defined as the proportion of patients being alive 12 months after their first administration of the study treatment (ipilimumab).
Efficacy according to immune-related response criteria (ir-RC) at any time during treatment | 12 months after date from the first study drug administration
Efficacy according RECIST criteria | 12 months after date from the first study drug administration
Progression free survival rate at 6 months | 6 months after date from the first study drug administration
Overall survival at 1 year in the subgroups (cutaneous, uveal, mucosal) | 12 months after date from the first study drug administration
To explore clinical efficacy of ipilimumab in relation to b-raf mutation status, brain metastases, LDH, HLA-A2 status | 12 months after date from the first study drug administration
To examine the value of peripheral blood absolute lymphocyte count (ALC) as a predictive biomarker in various patient cohorts with unresectable stage III-IV melanoma treated with ipilimumab monotherapy | 12 weeks after date from the first study drug administration
To evaluate possible surrogate markers in peripheral blood and tumour biopsy (translational research program) | 12 weeks after date from the first study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Schadendorf, Professor, Principal Investigator — University Hospital, Essen
Locations (25):
- Germany (25):
  - Universitätsklinikum Erlangen Hautklinik, Erlangen, Bavaria
  - Klinikum Nürnberg Nord, Nuremberg, Bavaria
  - Klinikum Kassel GmbH, Kassel, Hesse
  - Klinikum Dorothea Christiane Erxleben Quedlinburg gGmbH, Quedlinburg, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Universitätsklinikum Klinik f.Dermatologie, Allegologie u.Venerologie, Lübeck, Schleswig-Holstein
  - Charité Universitätsmedizin Berlin, Campus Mitte, Berlin
  - Krankenhaus Buxtehude, Buxtehude
  - Universitätsklinik Köln, Cologne
  - Helios Klinikum Erfurt, Erfurt
  - University Hospital Essen, Essen
  - Klinikum der Johann Wolfgang Goethe Universität, Frankfurt am Main
  - Universitätsklinikum Heidelberg Hautklinik, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg, Homburg/Saar
  - Klinik Universitätsklinikum Jena Klinik f. Hautkrankheiten, Jena
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Leipzig Dermatologie, Leipzig
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Mannheim gGmbH, Medizinische Fakultät Mannheim derUniversität Heidelberg, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - Ludwig-Maximilians-Universität München, München
  - Fachklinik Hornheide, Münster
  - Universitätsklinikum Münster Klinik u.Poliklinik f.Hautkrankheiten, Münster
  - Univ.-Klinikum Regensburg, Regensburg
  - Universitätshautklinik Tuebingen, Tübingen

REFERENCES:
- [Derived] Zimmer L, Eigentler TK, Kiecker F, Simon J, Utikal J, Mohr P, Berking C, Kampgen E, Dippel E, Stadler R, Hauschild A, Fluck M, Terheyden P, Rompel R, Loquai C, Assi Z, Garbe C, Schadendorf D. Open-label, multicenter, single-arm phase II DeCOG-study of ipilimumab in pretreated patients with different subtypes of metastatic melanoma. J Transl Med. 2015 Nov 6;13:351. doi: 10.1186/s12967-015-0716-5. PMID 26541511
- [Derived] Zimmer L, Vaubel J, Mohr P, Hauschild A, Utikal J, Simon J, Garbe C, Herbst R, Enk A, Kampgen E, Livingstone E, Bluhm L, Rompel R, Griewank KG, Fluck M, Schilling B, Schadendorf D. Phase II DeCOG-study of ipilimumab in pretreated and treatment-naive patients with metastatic uveal melanoma. PLoS One. 2015 Mar 11;10(3):e0118564. doi: 10.1371/journal.pone.0118564. eCollection 2015. PMID 25761109